CLINICAL TRIAL: NCT05215626
Title: Post-market Clinical Follow-up Study to Provide Safety, Performance and Clinical Benefits Data of the Zimmer® Reconstruction System (Implant and Instrumentation) - A Retrospective Consecutive Series Study
Brief Title: PMCF Study on the Safety, Performance and Clinical Benefits Data of the Zimmer® Reconstruction System
Status: Completed | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: MDRG2017-89MS-99T
Record Dates: First submitted 2022-01-28; First posted 2022-01-31 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Acetabulum Fracture; Pelvic Ring Fracture
Keywords: Acetabulum Fracture; Pelvic Ring Fracture; Medical Device; Clinical Benefits; Safety; Performance; Post Market Clinical Follow Up Study

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients implanted with the Zimmer Reconstruction System

SUMMARY:
The study is a monocentric, retrospective, non-randomized, non-controlled and consecutive series post-market study. The purpose of this study is to confirm safety, performance and clinical benefits of the Reconstruction System (implants and instrumentation) when used for temporary internal fixation and stabilization of fractures during the normal healing process.

The primary objective is the assessment of performance by analyzing fracture healing.

The secondary objectives are the assessment of safety by recording and analyzing the incidence and frequency of complications and adverse events. Relation of the events to implant, instrumentation and/or procedure should be specified. Subjects' outcomes will also be assessed.

DETAILED DESCRIPTION:
The Reconstruction System is especially used to stabilize pelvic ring and acetabulum fractures. One site will be involved in this study. The aim is to include a maximum of 83 consecutive series cases who received the Zimmer Reconstruction System at the Azienda Ospedaliero Universitaria Senese (Siena, Italy) between 2010 and 2018. All potential study subjects will be required to participate to the Informed Consent process.

Baseline data from the preop, intraop, immediate post-op and last consultation visit will be available in medical notes and collected retrospectively. In addition, any complications since the last consultation visit at the clinic and information about the treatment of the complications will also be collected retrospectively.

ELIGIBILITY:
Inclusion Criteria:

Patients having received the Zimmer Reconstruction System for temporary internal fixation and stabilization of fractures during the normal healing process

Exclusion Criteria:

* Off-label use
* Patients under the age of 18
* Severely comminuted fractures in which bone fragments are too small or numerous to adequately fix or maintain a reduced position
* Infection
* Metal sensitivity or intolerance
* Severe osteopenia and/or osteoporosis, or in the presence of marked or rapid bone absorption, metabolic bone disease, cancer, or any other tumor-like condition of the bone which may compromise fixation
* Sternal or spinal fractures
* Anatomical location in which the device would interfere with nerves, blood vessels, or other vital structures
* Patients with inadequate soft tissue coverage at the implant site

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive series of cases implanted with the Zimmer Reconstruction System according to Zimmer Biomet's Instruction for USE (IFU) and who meet the inclusion criteria and none of the exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-06-16 (Actual); Study Completion 2024-12-12 (Actual)

PRIMARY OUTCOMES:
Performance: Fracture healing | At last consultation visit at minimum 1 year postoperative.
  Performance will be assessed by analyzing fracture healing radiographically or clinically.

SECONDARY OUTCOMES:
Product safety | At operative evaluation, immediate post-operative evaluation and at last consultation visit at minimum 1 year postoperative.
  Safety will be assessed by recording and analyzing the incidence and frequency of complications and adverse events.
Harris Hip Score | At last consultation visit at minimum 1 year postoperative.
  Clinical benefits will be assessed by evaluating the Harris Hip Score (HHS). The HHS consists of four subscales (pain, function, the absence of deformity and range of motion). The survey has 10 question items and the score will range from 0 (worst) to 100 (best).

CONTACTS AND LOCATIONS:
Overall Officials: Hassan Achakri, Study Director — Zimmer Biomet
Locations (1):
- Azienda Ospedaliero Universitaria Senese, Siena, Italy